CLINICAL TRIAL: NCT00806234
Title: Improving Metabolic Parameters of Antipsychotic Child Treatment (IMPACT)
Brief Title: Reducing Weight Gain and Improving Metabolic Function in Children Being Treated With Antipsychotics
Acronym: IMPACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Maryland (Other); University of North Carolina, Chapel Hill (Other); The Zucker Hillside Hospital (Other)
Responsible Party: Principal Investigator, Mark Riddle, MD, Principal Investigator, Johns Hopkins University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH080270 (NIH); R01MH080270 (NIH); DSIR 84-CTS
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Psychotic Disorders
Keywords: Weight Gain; Obesity; IMPACT; Antipsychotic Treatment; Excessive Weight Gain Associated With Antipsychotic Treatment; Hybrid Efficacy/Effectiveness Design; Reducing Weight Gain; Improving Metabolic Parameters; Aripiprazole; Metformin; Risperdal; Seroquel; Quetiapine; Olanzapine; Zyprexa; Geodon; Risperidone; Abilify; Trilafon; Perphenazine; Glucophage; Paliperidone; Olanzapine/fluoxetine
MeSH Terms: conditions — Psychotic Disorders; Weight Gain; Obesity; Tooth, Impacted | interventions — Aripiprazole; Perphenazine; Metformin; Olanzapine; Quetiapine Fumarate; Risperidone; ziprasidone; asenapine; iloperidone; Lurasidone Hydrochloride; Paliperidone Palmitate; Fluoxetine; olanzapine-fluoxetine combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Participants will continue on current antipsychotic medication.
  Interventions: Drug: Olanzapine, quetiapine, risperidone, ziprasidone, aripiprazole, asenapine, iloperidone, lurasidone, paliperidone, or olanzapine/fluoxetine
- 2 (Experimental): Participants will undergo a staggered switch from current antipsychotic medication to aripiprazole or perphenazine.
  Interventions: Drug: Aripiprazole or Perphenazine
- 3 (Experimental): Participants will add metformin to current antipsychotic medication treatment.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Aripiprazole or Perphenazine — Baseline second generation antipsychotic (SGA) treatment will be gradually decreased and discontinued over 8 weeks while treatment with aripiprazole or perphenazine will be increased to effective levels.
  Other Names: Abilify, Trilafon
  Arms: 2
Drug: Metformin — Metformin treatment will be added to current SGA treatment, with dosing based on participant weight and increased according to a preset titration schedule unless side effects interfere.
  Other Names: Glucophage
  Arms: 3
Drug: Olanzapine, quetiapine, risperidone, ziprasidone, aripiprazole, asenapine, iloperidone, lurasidone, paliperidone, or olanzapine/fluoxetine — Current antipsychotic medication will be continued throughout the treatment period, with changes in dose only made as clinically indicated
  Other Names: Zyprexa, Seroquel, Risperdal, Geodon, Abilify, Saphris, Sycrest, Fanapt, Fanapta, Zomaril, Latuda, Invega, Symbyax
  Arms: 1

SUMMARY:
This study will test the effectiveness of two different treatments for children and adolescents who have gained weight on their antipsychotic medications.

DETAILED DESCRIPTION:
Disorders that involve severe dysregulation of mood or thoughts in children -- such as early onset bipolar spectrum (BPS) and schizophrenia spectrum (SS) disorders -- are commonly treated with antipsychotic medications. However, many of the newest and most commonly prescribed antipsychotic medications can cause weight gain and metabolic dysfunctions. Use of these newer antipsychotics, called second generation antipsychotics (SGAs), is increasing rapidly in children, and the risk of weight gain from SGAs is higher among children than adults. Excessive weight gain can lead to obesity, which, in turn, can lead to increased health care costs, increased risk of sickness, and lower life expectancy. These factors are enhanced in children and adolescents who grow up obese.

Two different strategies to reduce weight gain and metabolic side effects from SGAs will be tested in this study. The first strategy involves switching from the current SGA to a lower risk agent (aripiprazole or perphenazine) hypothesized to result in weight loss and improved metabolic functioning. The second strategy involves taking the medication metformin in addition to the current SGA. Metformin is approved by the Food and Drug Administration (FDA) to promote weight loss in youth with diabetes and has been effective in reducing weight in youth taking SGAs.

Participation in this study will last between 26 and 27 weeks and will be divided into two parts. The first part will last 2 to 3 weeks and include three study visits. During this part, participants will undergo a physical exam, an electrocardiogram (EKG), a dual energy X-ray absorptiometry (DXA) test, and blood tests. The DXA measures body fat.

The second part will last 24 weeks and include nine study visits. During this part, participants will be randomly assigned to one of three conditions: gradual switch of current SGA medication to either aripiprazole or perphenazine, addition of metformin to current SGA medication, or no change to treatment with current SGA medication. Visits will take place on Weeks 1, 2, 4, 6, 8, 12, 16, 20, and 24. At each visit, participants will meet with a study doctor who will assess symptoms and side effects, and participants and their guardians will receive information and recommendations about childhood obesity and weight loss. There will also be monthly urine pregnancy tests, and two blood tests.

ELIGIBILITY:
Inclusion Criteria:

* DSM diagnoses that have an FDA indication for atypical antipsychotic use for at least one agent in the respective pediatric or adult age group. Specifically, primary DSM-IV diagnosis of Early Onset Schizophrenia Spectrum (EOSS; schizophrenia, schizoaffective disorder, schizophreniform disorder, psychotic disorder NOS); Bipolar Spectrum (bipolar I, II and NOS); Major depressive disorder with psychosis; Mood disorder NOS corresponding to Leibenluft and colleagues severely mood dysregulated (SMD) broad spectrum bipolar disorder; Mood disorder NOS corresponding to irritability associated with autism spectrum disorders; or - for adult teen participants aged 18-19 years - Major depressive disorder. Diagnoses will be determined by clinical interview, Leibenluft's modification of the K-SADS-PL, and the "Aberrant Behavior Checklist" (cutoff score of 18, as used by FDA for approval of risperidone and aripiprazole in minors).
* Clinically stable on current treatment regimen for at least 30 days, as assessed in a three-step process
* Current SGA treatment with olanzapine, quetiapine, risperidone, ziprasidone aripiprazole, asenapine, iloperidone, lurasidone, paliperidone, or olanzapine/fluoxetine for ≥ 8 weeks
* Stable dose of current SGA and psychotropic co-medications for at least 30 days
* Body mass index (BMI) at least in the 85th percentile for age and gender
* Substantial weight gain over the previous 3 years while taking a SGA, as reflected by family and referring physician's judgment. The weight gain did not have to occur on the child's current SGA. Weight needs to have remained stable or increased over past year.
* Agrees to use two effective forms of birth control or to remain abstinent
* Has a primary caretaker who has known the child well for at least 6 months before study entry
* Primary caretaker is able to participate in study appointments as clinically indicated

Exclusion Criteria:

* Treatment with any medication (other than the currently prescribed psychotropic medications) that would significantly alter glucose, insulin, or lipid levels. Exception: orlistat and amantadine are permitted if the individual has taken the drug for at least one year without weight loss.
* Major neurological or medical illness that affects weight gain or that would prevent participation in physical activities
* Fasting glucose levels indicating need for prompt treatment
* Pediatrician or pediatric gastroenterologist recommendation to address abnormal fasting labs by pursuing more active treatment than those in the 2007 American Medical Association guidelines
* Diagnosis of anorexia nervosa or bulimia nervosa, as based on current or lifetime DSM-IV criteria
* Diagnosis of substance dependence disorder (other than tobacco dependence) within the past month, as based on DSM-IV criteria
* Positive urine toxicology indicating ongoing use of illicit substance
* Current treatment with more than one antipsychotic medication
* Current treatment with more than 3 total psychotropic medications (i.e., 2 psychotropics plus SGA), with the exception of subjects taking 2 medications for ADHD in which a total of 4 psychotropic medications are allowed.
* Known hypersensitivity to metformin
* Prior treatment with aripiprazole and perphenazine for more than 2 weeks that was stopped for inefficacy or intolerability
* Pregnant, breastfeeding, or unwilling to comply with contraceptive requirements of study
* IQ score less than 55
* Significant risk of dangerousness to self or to others that would make study participation inadvisable
* Language issues that prevent child and/or parent from completing assessments or treatment
* Ongoing or previously undisclosed child abuse requiring new department of social service intervention

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 127 (Actual)
Dates: Start 2009-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Reeves, MD, Principal Investigator — University of Maryland; Linmarie Sikich, MD, Principal Investigator — University of North Carolina, Division of Child and Adolescent Psychiatry; Christoph Correll, MD, Principal Investigator — The Zucker Hillside Hospital; Mark A. Riddle, MD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - University of North Carolina, Division of Child and Adolescent Psychiatry, Chapel Hill, North Carolina

REFERENCES:
- [Background] Reeves GM, Keeton C, Correll CU, Johnson JL, Hamer RM, Sikich L, Hazzard L, Alderman C, Scheer A, Mabe M, Kapoor S, Sheridan E, Borner I, Bussell K, Pirmohamed S, Bethea TC, Chekuri R, Gottfried R, Reinblatt SP, Santana E, Riddle MA. Improving metabolic parameters of antipsychotic child treatment (IMPACT) study: rationale, design, and methods. Child Adolesc Psychiatry Ment Health. 2013 Aug 15;7(1):31. doi: 10.1186/1753-2000-7-31. PMID 23947389

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Lifestyle Information: Participants will continue on current antipsychotic medication.
  Olanzapine, quetiapine, risperidone, ziprasidone, aripiprazole, asenapine, iloperidone, lurasidone, paliperidone, or olanzapine/fluoxetine: Current antipsychotic medication will be continued throughout the treatment period, with changes in dose only made as clinically indicated
- Switch Treatment + Healthy Lifestyle Instruction: Participants will undergo a staggered switch from current antipsychotic medication to aripiprazole or perphenazine.
  Aripiprazole or Perphenazine: Baseline second generation antipsychotic (SGA) treatment will be gradually decreased and discontinued over 8 weeks while treatment with aripiprazole or perphenazine will be increased to effective levels.
- Metformin Treatment + Healthy Lifestyle Instruction: Participants will add metformin to current antipsychotic medication treatment.
  Metformin: Metformin treatment will be added to current SGA treatment, with dosing based on participant weight and increased according to a preset titration schedule unless side effects interfere.
Period: Overall Study
Arm/Group | Healthy Lifestyle Information | Switch Treatment + Healthy Lifestyle Instruction | Metformin Treatment + Healthy Lifestyle Instruction
Started | 47 | 31 | 49
Completed | 34 | 19 | 37
Not Completed | 13 | 12 | 12

BASELINE CHARACTERISTICS:
Population: 127 subjects were randomized between 10/2009-10/2013 into three groups (CONTROL=47; MET=49; SWITCH=31). Safety analyses excluded 4 participants (CONTROL=1, MET=2, SWITCH=1) who discontinued at baseline. Primary efficacy analyses included 121 participants (CONTROL=44; MET=47; SWITCH=30) with ≥1 post-baseline vital sign measurement.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Lifestyle Information | Switch Treatment + Healthy Lifestyle Instruction | Metformin Treatment + Healthy Lifestyle Instruction | Total
Number analyzed (Participants) | 47 | 31 | 49 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41 | 26 | 45 | 112
  Between 18 and 65 years | 6 | 5 | 4 | 15
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 18 | 45
  Male | 30 | 21 | 31 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 7 | 16
  Not Hispanic or Latino | 42 | 27 | 42 | 111
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 9 | 14 | 36
  White | 25 | 16 | 26 | 67
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 6 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (BMI) Z-score Change
Time Frame: Change from baseline to 24 weeks
Measure: Least Squares Mean (Standard Error); unit: Z Score
Arm/Group | Healthy Lifestyle Information | Switch Treatment + Healthy Lifestyle Instruction | Metformin Treatment + Healthy Lifestyle Instruction
Number analyzed (Participants) | 44 | 30 | 47
Z Score | 0.040 (0.029) | -0.112 (0.037) | -0.088 (0.028)

2. Secondary Outcome: Change in Whole Body Insulin Sensitivity Index
Time Frame: Change from baseline to 24 weeks
Measure: Least Squares Mean (Standard Error); unit: mU/L
Arm/Group | Healthy Lifestyle Information | Switch Treatment + Healthy Lifestyle Instruction | Metformin Treatment + Healthy Lifestyle Instruction
Number analyzed (Participants) | 44 | 30 | 47
mU/L | 0.74 (0.82) | 0.42 (0.91) | -0.34 (0.65)

3. Secondary Outcome: Triglyceride Levels
Time Frame: Change from baseline to 24 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Healthy Lifestyle Information | Switch Treatment + Healthy Lifestyle Instruction | Metformin Treatment + Healthy Lifestyle Instruction
Number analyzed (Participants) | 44 | 30 | 47
mg/dL | 0.2 (9.1) | 16.6 (12.0) | 14.7 (8.7)

4. Secondary Outcome: Change in Low Density Lipoprotein (LDL) Cholesterol Level
Time Frame: From Baseline to Week 24
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Healthy Lifestyle Information | Switch Treatment + Healthy Lifestyle Instruction | Metformin Treatment + Healthy Lifestyle Instruction
Number analyzed (Participants) | 44 | 30 | 47
mg/dL | 3.6 (4.2) | -8.1 (5.4) | -4.1 (3.9)

ADVERSE EVENTS:
Description: See the correct numbers for the 3 populations below. We had to exclude 5 participants (CONTROL = 2, METFORMIN = 2, SWITCH = 1).
  1. Randomized population:
     Control - 47 Metformin - 49 Switch - 31
     Aripiprazole - 13 Molindone - 1 Perphenazine - 17
  2. Safety population:
     Control - 45 Metformin - 47 Switch - 30
     Aripiprazole - 12 Molindone - 1 Perphenazine - 17
  3. Efficacy population :
  Control - 44 Metformin - 47 Switch - 30
  Aripiprazole - 12 Molindone - 1 Perphenazine - 17
Arm/Group | Healthy Lifestyle Information | Switch Treatment + Healthy Lifestyle Instruction | Metformin Treatment + Healthy Lifestyle Instruction
Serious Adverse Events (participants affected / at risk) | 1/45 | 5/30 | 3/47
Other Adverse Events (participants affected / at risk) | 45/45 | 30/30 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Lifestyle Information (N=45) | Switch Treatment + Healthy Lifestyle Instruction (N=30) | Metformin Treatment + Healthy Lifestyle Instruction (N=47)
Femur Fracture (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Asthma attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Lifestyle Information (N=45) | Switch Treatment + Healthy Lifestyle Instruction (N=30) | Metformin Treatment + Healthy Lifestyle Instruction (N=47)
Abdominal pain or discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
Agitation (Nervous system disorders) | 8 (8) | 6 (6) | 5 (5)
Hypersomnia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Aggression or hostility (Psychiatric disorders) | 10 (10) | 6 (6) | 3 (3)
Anger or irritability (Psychiatric disorders) | 9 (9) | 6 (6) | 5 (5)
Impulse-control disorder (Psychiatric disorders) | 4 (4) | 4 (4) | 1 (1)
Negativism (Psychiatric disorders) | 4 (4) | 5 (5) | 6 (6)
Frustration (Psychiatric disorders) | 4 (4) | 4 (4) | 4 (4)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 6 (6)
Mood swings (Psychiatric disorders) | 2 (2) | 2 (2) | 4 (4)
Obsessive rumination (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Infection (General disorders) | 4 (4) | 3 (3) | 8 (8)
Acne (General disorders) | 1 (1) | 2 (2) | 0 (0)
Energy increased (General disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting or nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Restlessness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Initial Insomnia (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Injury (General disorders) | 3 (3) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Depressed Mood (Psychiatric disorders) | 4 (4) | 2 (2) | 1 (1)
Hallucination (Psychiatric disorders) | 4 (4) | 1 (1) | 2 (2)
Disturbance in attention (Psychiatric disorders) | 3 (3) | 0 (0) | 4 (4)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2)
Psychomotor hyperactivity (Psychiatric disorders) | 2 (2) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
27 subjects were randomized between 10/2009-10/2013 into three groups (CONTROL=47; MET=49; SWITCH=31). Safety analyses excluded 4 participants (CONTROL=1, MET=2, SWITCH=1) who discontinued at baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No